CLINICAL TRIAL: NCT00788008
Title: Does Inhalational Anesthesia Accelerate Postoperative Cognitive Decline?
Brief Title: Cognitive Effects of Inhalational Versus Intravenous General Anesthesia in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00010070
Record Dates: First submitted 2008-11-06; First posted 2008-11-10 (Estimated); Results first posted 2015-03-26 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Lumbar Spondylosis; Cervical Spondylosis; Hip Osteoarthritis; Knee Osteoarthritis
Keywords: spinal, joint
MeSH Terms: conditions — Spondylosis; Osteoarthritis, Hip; Osteoarthritis, Knee | interventions — Anesthesia, Inhalation; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Inhalational anesthesia with isoflurane
  Interventions: Drug: inhalation anesthesia with isoflurane vs. TIVA with propofol
- 2 (Active Comparator): total intravenous anesthesia with propofol
  Interventions: Drug: inhalation anesthesia with isoflurane vs. TIVA with propofol

INTERVENTIONS:
Drug: inhalation anesthesia with isoflurane vs. TIVA with propofol — variable depending upon patient
  Other Names: Diprivan

SUMMARY:
The purpose of this research is to determine if post-operative cognition will be better if the general anesthesia for surgery is done with an inhaled (gas through a breathing tube) or intravenous (medicine injected in the IV) general anesthetic technique.

DETAILED DESCRIPTION:
A prospective randomized pre-test post-test design will be used. After obtaining informed consent, patients will be randomized to either: 1) Inhalational anesthesia with isoflurane or 2) Total intravenous anesthesia(TIVA) with propofol. Randomization will be stratified by surgical type so that this variable is equally distributed between the treatment groups. All patients will be maintained at a standard depth of anesthesia (40-60) using a Bispectral Index (BIS®) monitor. Normocarbia will be maintained in the operating room using capnography monitoring. Normothermia will be maintained throughout the procedure.

The anesthesia team providing care for these patients will be able to choose the premedication and muscle relaxant for the anesthetic technique. Patient controlled anesthesia or regional anesthetic techniques may be used for post-operative analgesia at the discretion of the anesthesia team providing care for these patients. Anesthesia will be induced with intravenous propofol and fentanyl in all patients, unless contraindicated. Patients will be mechanically ventilated with air/oxygen. Temperature will be maintained > 35º C and ventilation will be adjusted to maintain end-tidal carbon dioxide (CO2) at 35 ± 5 mmHg. Mean arterial pressure will be maintained ≥ 75% of baseline or ≥ 60 mmHg, whichever is greater, in both groups. After induction of anesthesia, the maintenance anesthesia will consist of either:

1. Inhalational anesthesia group - isoflurane will be used for maintenance of anesthesia. Intravenous fentanyl and/or remifentanil will be used for supplementary analgesia. These agents will be administered to maintain a normal depth of anesthesia using the BIS® monitor and traditional signs of anesthetic depth.
2. TIVA group - propofol and opioid infusions (fentanyl or remifentanil) will be used for the maintenance of anesthesia. The infusions will be adjusted to maintain a normal depth of anesthesia using the BIS® monitor along with traditional signs of anesthetic depth.

All subjects will undergo pre-operative neurocognitive testing within two weeks of their surgery, and at 3 months post-surgery. The persistence versus resolution of cognitive deficits over time will be determined with a 1 year post-surgical follow-up assessment. Pre- to post-test change scores will be compared across groups on primary and secondary outcome variables (see below) while controlling for relevant demographic variables (age, education, sex).

ELIGIBILITY:
Inclusion Criteria:

* patients (aged 65 years or older) scheduled for elective spine or major joint replacement (total hip or total knee arthroplasty) at Duke University Medical Center or the Durham VA Medical Center

Exclusion Criteria:

* not fluent in English and able to comprehend the English language
* have severe visual or auditory handicaps
* Carry a diagnosis of dementia or score < 18 on the Mini-Mental State Examination (MMSE) as calculated from the Modified Mini-Mental State (3MS) (see D4 below)
* have allergies to eggs, propofol, isoflurane, fentanyl, remifentanil, or pregabalin

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terri G Monk, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - VAMC, Durham, North Carolina

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 200 patients were consented. One person dropped out prior to baseline testing.
Groups:
- Isoflurane: Inhalational anesthesia with isoflurane
- Propofol: Total intravenous anesthesia with propofol
Period: Overall Study
Arm/Group | Isoflurane | Propofol
Started | 98 | 101
Completed | 98 | 101
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Isoflurane | Propofol | Total
Number analyzed (Participants) | 98 | 101 | 199
Age, Continuous [Mean (Full Range); unit: years] | 73.38 [66 to 86] | 73.13 [65 to 91] | 73.25 [65 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 39 | 71
  Male | 66 | 62 | 128
Region of Enrollment [Number; unit: participants]
  United States | 98 | 101 | 199

OUTCOME MEASURES:

1. Primary Outcome: Change in Neurocognitive Performance (Z-score)
Description: Mean change on composite scores (z-score) for memory and executive function measures.
  Memory measures: Hopkins Verbal Learning Test-Revised and the Brief Visuospatial Memory Test-Revised.
  Executive function measures: the Trail Making Test (Army, 1944), Digit-symbol substitution and Symbol Search subtests of the Processing Speed Index of the Wechsler Adult Intelligence Scale-III (WAIS-III; Wechsler, 1997) and the Controlled Oral Word Association subtest of the Multilingual Aphasia Examination.
  The outcomes were constructed as summed z-score composites. They are scaled as standard deviations. Thus, a score of 0 was central on each composite, and 95% of the scores would fall within -2.0 and +2.0. While there is no minimum or maximum value is rare for any score (<1%) to fall outside the -3.0 to +3.0 range.
  Higher scores (and thus positive change value) indicate an improvement of function.
Time Frame: 3 months post operatively
Measure: Mean (Full Range); unit: z score
Arm/Group | Isoflurane | Propofol
Number analyzed (Participants) | 98 | 101
z score
  Memory measures | .09 [-3.3 to 3.3] | -.20 [-3.3 to 3.3]
  Executive Function measures | -.42 [-8.0 to 4.4] | .01 [-8.0 to 4.4]

ADVERSE EVENTS:
Description: Only unexpected adverse events that were related to the study were collected.
Arm/Group | Isoflurane | Propofol
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/101
Other Adverse Events (participants affected / at risk) | 0/98 | 0/101

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No